CLINICAL TRIAL: NCT00530790
Title: Clinical Evaluation of Ropinirole CR-RLS Tablets in Restless Legs Syndrome-Open-Label, Uncontrolled Study. Classification: Clinical Pharmacology, Exploratory
Brief Title: Clinical Evaluation of Ropinirole CR-RLS ( SK&F101468)Tablets in Restless Legs Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107846
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Results first posted 2009-07-24 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

ARMS (1):
- ropinirole CR-RLS (Experimental): Subjects will orally take ropinirole CR-RLS tablet(s) once daily 1-2 hours before the onset of RLS symptoms at about the same time of the day. The time of taking ropinirole must be after 16:00.Adjustment of the Ropinirole CR-RLS tablets should be completed after the Week 1 visit up to the Week 10 visit. The dose will be increased at intervals of at least one week until sufficient efficacy is obtained (use "much improved" as a guide) without safety problem. Dose escalation will start at the initial dose 0.5 mg/day to 1 mg/day; after 1 mg/day, the dose will be increased by 1 mg/day to the maximum 6 mg/day.
  Interventions: Drug: ropinirole controlled release (CR)-RLS

INTERVENTIONS:
Drug: ropinirole controlled release (CR)-RLS — White film-coated round-shaped tablet
  Other Names: Ropinirole CR-RLS (SK&F101468)

SUMMARY:
This study was designed to evaluate the safety, pharmacokinetic profile and efficacy in Restless Legs Syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be considered eligible for inclusion in this study only if all of the following criteria apply:

At Week -1 (at the start of Screening period)

* Patients who are diagnosed with RLS according to the International RLS Study Group's (IRLSSG) Diagnostic Criteria.
* Age: Patients aged at least 18 years and under 80 years.
* Patients who have had RLS symptoms in the evening or nighttime (17:00 to 7:00 next day) for at least 20 days within one month before the start of the screening period. Patients treated for RLS before the start of the Screening period and who do not meet this criterion are considered eligible if the previous therapy can be discontinued from the Screening period.
* Patients who experience RLS symptoms requiring treatment after 17:00 but prior to bedtime.
* Gender: male and female Female of child-bearing potential will be eligible for inclusion in this study. However they must have a negative pregnancy test at the Screening visit. They agree are perform pregnancy test at the time determined and practice one of the following method of contraception from the Screening visit till the end of follow-up examination.

  * Abstinence
  * Oral Contraceptive, either combined or progestogen alone
  * Injectable progestogen
  * Implants of levonorgestrel
  * Estrogenic vaginal ring
  * Percutaneous contraceptive patches
  * Intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label
  * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
  * Double barrier method: condom or occlusive cap (diaphragm or cervical / vault caps) plus spermicidal agent (foam /gel / film / cream / suppository
* Inpatient or outpatient status: Outpatient status
* Patients who are able to give informed written consent in person. For patients aged under 20 years, their legally acceptable representatives are able to give informed written consent.

At Week 0 (at the start of treatment period)

* Patients who experience RLS symptoms in the evening and nighttime (17:00 to 7:00 next day) for at least 4 days within 7 days before the start of the treatment period.
* Patients who have sleep impairment associated with RLS. Patients who answered as 3 (severe) or 4 (very severe) to Question 4 (Sleep disturbance) in the IRLS Rating Scale
* Patients whose IRLS Rating Scale total scores are 15 points or more.

Exclusion Criteria:

* Patients requiring treatment for daytime RLS symptoms (7:00 to 17:00).
* Patients with signs of secondary RLS (e.g. chronic renal failure, iron-deficiency anemia, pregnancy, rheumatoid arthritis and Parkinson's disease).
* Patients whose serum ferritin level is <10 μg/L (ng/mL) at the start of Screening period.
* Patients with following sleep disorder not associated with RLS e.g. narcolepsy, sleep terror disorder, sleep walking disorder, breathing related sleep disorder (Patients with obvious apnea in nighttime sleeping when they do not have alcohol drinking or over 15 times/hour is used to a target for apnea hypopnea index,in which case to implement polysomnography), etc.
* Patients with complication of movement disorder (e.g. Parkinson's disease, dyskinesia, dystonia, etc.).
* Patients with severe hepatic/renal/cardiac/pulmonary disorder or hematopoietic disorder.

The severity refers to Grade 3 according to "the Classification of the Severity of Adverse Experiences" (Pharmaceutical affairs Bureau/Safety Division (PAB/SD) Notification No. 80, dated 29 June 1992).

* Patients with the medical history or complication of cancer or malignant tumour.
* Patients with the medical history or complication of substance abuse (e.g. alcohol or drug) or dependency of substance for the last one year
* Patients whose diastolic blood pressure (BP) is >110 mmHg or <50 mmHg or whose systolic BP is >180 mmHg or <90 mmHg at the start of Screening period and Week0.
* Patients intolerant for ropinirole hydrochloride (HCl) or other dopamine agonists.
* Patients with the medical history of allergy to ropinirole HCl in the past.
* Patients with the medical history of Augmentation to ropinirole HCl or other dopamine agonists in the past and those who have experienced early morning RLS symptoms.

Augmentation is defined as below:

RLS appear 2 hours earlier than the pre-treatment. Symptoms become severer than the pre-treatment. Symptoms which start after less time at rest than they did before treatment. The RLS extend to other sites (e.g. arm and trunk).

* Patients without nighttime sleeping habit (e.g. night-shift worker, etc.) and those who must drastically change the habitual bedtime during the study duration.
* Patients who have participated in another clinical study of an investigational product or medical device within the last 12 weeks prior to the start of screening period.
* Female patients who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study .
* Patients with chronic hepatitis typeB and /or typeC which is positive of hepatitis B surface antigen （HBsAg）and/or hepatitis C antibody.
* Patients who have medical conditions which, in the opinion of investigator could affect efficacy and safety assessment. This may include, but are not limited to the following disorders: diabetes, peripheral neuropathy, fibromyalgia syndrome, symptomatic orthostatic hypotension, hepatic or renal failure, pleuro-pulmonary fibrosis.
* Patients who have received treatment of an estrogen drug product and a drug that are known to substantially inhibit CYP1A2 and have changed the dose from baseline visit to Week 0.
* Others whom the investigator (sub investigator) considers ineligible for the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-08-23; Primary Completion 2008-02-01 (Actual); Study Completion 2008-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Japan (6):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] GSK has concluded that it is not feasible to publish this study in a peer-reviewed scientific journal because the nature of the study is unlikely to be of interest to a journal. GSK is providing the attached study results summary with a conclusion.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 107846 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107846 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107846 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107846 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Ropinirole CR-RLS: Subjects who took oral Ropinirole CR-RLS once daily 1-2 hours before onset of Restless Legs Syndrome (RLS) symptoms (after 4pm). Initial dose level was 0.5 mg/day and increased weekly by 1 mg/day until sufficient efficacy was obtained without any tolerability issues. Treatment period was 12 weeks. Maximum dose level was 6 mg per day.
Period: Overall Study
Arm/Group | Ropinirole CR-RLS
Started | 35
Completed | 30
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 12
Region of Enrollment [Number; unit: Number of participants]
  Japan | 35

OUTCOME MEASURES:

1. Primary Outcome: Drug Related Adverse Events-On-Therapy
Time Frame: Weeks 1 - 12 Treatment Period
Population: Safety Population consisting of the subjects who took at least one dose of the study medication.
Measure: Number; unit: Number of Events
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Number of Events
  Subjects with any Adverse Events | 29
  Nausea | 14
  Somnolence | 5
  Vomiting | 5
  Hypersomnia | 3
  Diarrhea | 2
  Dizziness | 2
  Dyspepsia | 2
  Fatigue | 2
  Stomach discomfort | 2
  Abdominal pain | 1
  Anemia | 1
  Insomnia | 1
  Irritability | 1
  Malaise | 1
  Middle Insomnia | 1
  Motion Sickness | 1
  Palpitations | 1
  Thirst | 1

2. Secondary Outcome: Change From Baseline to Week 12 in International Restless Leg Syndrome (IRLS) Rating Scale Total Score
Description: The IRLS Scale assesses the severity of sensory and motor symptoms, sleep disturbance, daytime somnolence, and impact on activities of daily living and mood. The questionnaire scores various questions and totals them using the following scale: Very severe=31-40 points, Severe=21-30 points, Moderate=11-20 points, Mild=1-10 points, None=0 points.
Time Frame: Baseline and after Week 12
Population: Full Analysis Set: Subjects entered to the treatment period, except for those not fulfilling the major registration criteria, those who did not take even one dose of the study medication, and those for whom no observation data were available after starting the study treatment. Method for missing data is Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Points on a scale
  IRLS assessment Score - week 0 | 25.3 (4.42)
  IRLS assessment Score - week 12 | 6.0 (7.5)
  Change from Baseline at week 12 | -19.3 (7.68)

3. Secondary Outcome: Clinical Global Impression Scale - Severity of Illness (CGI-S)
Description: The CGI-S scale measures the overall severity of illness on a 7 point scale. Normal = 1, Borderline = 2, Mildly = 3, Moderately = 4, Markedly = 5, Severely = 6, Extremely Severe = 7(no subjects scored a 7).
Time Frame: Baseline - Final assessment point
Population: Full Analysis Set Population (Baseline, Weeks 1, 2, 3, 4 = 35 subjects; Weeks 5 and 6 = 33 subjects; Week 8 = 32 subjects; Weeks 10 and 12 = 30 subjects; Final assessment point = 35 subjects). Method of Missing Data = LOCF.
Measure: Number; unit: Participants
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Participants
  Baseline - Normal | 0
  Baseline - Borderline | 0
  Baseline - Mildly | 0
  Baseline - Moderately | 13
  Baseline - Markedly | 13
  Baseline - Severely | 9
  Week 1 - Normal | 0
  Week 1 - Borderline | 3
  Week 1 - Mildly | 10
  Week 1 - Moderately | 16
  Week 1 - Markedly | 4
  Week 1 - Severely | 2
  Week 2 - Normal | 3
  Week 2 - Borderline | 7
  Week 2 - Mildly | 12
  Week 2 - Moderately | 10
  Week 2 - Markedly | 2
  Week 2 - Severely | 1
  Week 3 - Normal | 11
  Week 3 - Borderline | 7
  Week 3 - Mildly | 8
  Week 3 - Moderately | 7
  Week 3 - Markedly | 1
  Week 3 - Severely | 1
  Week 4 - Normal | 9
  Week 4 - Borderline | 9
  Week 4 - Mildly | 10
  Week 4 - Moderately | 5
  Week 4 - Markedly | 1
  Week 4 - Severely | 1
  Week 5 - Normal | 11
  Week 5 - Borderline | 6
  Week 5 - Mildly | 11
  Week 5 - Moderately | 4
  Week 5 - Markedly | 1
  Week 5 - Severely | 0
  Week 6 - Normal | 13
  Week 6 - Borderline | 4
  Week 6 - Mildly | 11
  Week 6 - Moderately | 4
  Week 6 - Markedly | 1
  Week 6 - Severely | 0
  Week 8 - Normal | 10
  Week 8 - Borderline | 10
  Week 8 - Mildly | 8
  Week 8 - Moderately | 3
  Week 8 - Markedly | 1
  Week 8 - Severely | 0
  Week 10 - Normal | 15
  Week 10 - Borderline | 5
  Week 10 - Mildly | 8
  Week 10 - Moderately | 1
  Week 10 - Markedly | 1
  Week 10 - Severely | 0
  Week 12 - Normal | 16
  Week 12 - Borderline | 3
  Week 12 - Mildly | 10
  Week 12 - Moderately | 0
  Week 12 - Markedly | 1
  Week 12 - Severely | 0
  Final assessment point - Normal | 17
  Final assessment point - Borderline | 3
  Final assessment point - Mildly | 12
  Final assessment point - Moderately | 1
  Final assessment point - Markedly | 1
  Final assessment point - Severely | 1

4. Secondary Outcome: Clinical Global Impression Global Improvement (CGI-GI)
Description: CGI-GI is a 7 point scale assessing Global Improvement. 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse (no patients scored a 5, 6, or 7).
Time Frame: Baseline - Final assessment point
Population: Full Analysis Set Population (Weeks 1, 2, 3, and 4 = 35 subjects; Weeks 5 and 6 = 33 subjects; Week 8 = 32 subjects; Week 10, 12 = 30 subjects; Final assessment point = 35 subjects). Method for missing date is LOCF.
Measure: Number; unit: Participants
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Participants
  Week 1 - Very Much Improved | 4
  Week 1 - Much Improved | 12
  Week 1 - Minimally Improved | 13
  Week 1 - No Change | 6
  Week 2 - Very Much Improved | 15
  Week 2 - Much Improved | 9
  Week 2 - Minimally Improved | 9
  Week 2 - No Change | 2
  Week 3 - Very Much Improved | 21
  Week 3 - Much Improved | 7
  Week 3 - Minimally Improved | 6
  Week 3 - No Change | 1
  Week 4 - Very Much Improved | 21
  Week 4 - Much Improved | 7
  Week 4 - Minimally Improved | 6
  Week 4 - No Change | 1
  Week 5 - Very Much Improved | 21
  Week 5 - Much Improved | 6
  Week 5 - Minimally Improved | 6
  Week 5 - No Change | 0
  Week 6 - Very Much Improved | 22
  Week 6 - Much Improved | 7
  Week 6 - Minimally Improved | 4
  Week 6 - No Change | 0
  Week 8 - Very Much Improved | 24
  Week 8 - Much Improved | 6
  Week 8 - Minimally Improved | 2
  Week 8 - No Change | 0
  Week 10 - Very Much Improved | 22
  Week 10 - Much Improved | 6
  Week 10 - Minimally Improved | 2
  Week 10 - No Change | 0
  Week 12 - Very Much Improved | 25
  Week 12 - Much Improved | 4
  Week 12 - Minimally Improved | 0
  Week 12 - No Change | 1
  Final assessment point - Very Much Improved | 27
  Final assessment point - Much Improved | 5
  Final assessment point - Minimally Improved | 1
  Final assessment point - No Change | 2

5. Secondary Outcome: Change From Baseline at Week 12/Early Withdrawal (EW) in Pittsburgh Sleep Quality Index (PSQI) Total Score
Description: The PSQI generates seven scores that correspond to different domains. Each component score ranges from 0 (no difficulty) to 3 (severe difficulty). The domain scores are totaled to produce a global score (range of 0-21). A PSQI global score > 5 is considered to be suggestive of significant sleep disturbance.
Time Frame: Baseline - Week 12/EW
Population: Full Analysis Set(FAS)
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Points on a scale
  PSQI Total Score at Baseline | 9.4 (3.20)
  PSQI Total Score at Week 12/EW | 5.4 (2.89)
  Change from Baseline at Week 12/EW | -4.2 (3.94)

6. Secondary Outcome: Change From Baseline to Week 12/EW in Pittsburgh Sleep Quality Index (PSQI) Total Score by Domains
Description: as for outcome 5
Time Frame: Baseline - Week 12/EW
Population: Full Analysis Set(FAS)
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Points on a scale
  Sleep Quality - Baseline | 2.0 (0.62)
  Sleep Quality - Week 12/EW | 1.2 (0.77)
  Sleep Quality - Change from Baseline | -0.9 (0.78)
  Duration getting to sleep - Baseline | 2.0 (1.04)
  Duration getting to sleep - Week 12/EW | 1.0 (0.88)
  Duration getting to sleep - Change from Baseline | -1.1 (1.09)
  Sleep Duration - Baseline | 1.9 (0.77)
  Sleep Duration - Week 12/EW | 1.5 (0.79)
  Sleep Duration - Change from Baseline | -0.4 (0.74)
  Sleep Adequacy - Baseline | 0.9 (1.11)
  Sleep Adequacy - Week 12/EW | 0.4 (0.70)
  Sleep Adequacy - Change from Baseline | -0.6 (1.19)
  Sleep Disturbance - Baseline | 1.2 (0.43)
  Sleep Disturbance - Week 12/EW | 0.9 (0.55)
  Sleep Disturbance - Change from Baseline | -0.3 (0.60)
  Use of Sleeping pill - Baseline | 0.4 (1.01)
  Use of Sleeping pill - Week 12/EW | 0.0 (0.00)
  Use of Sleeping pill - Change from Baseline | -0.4 (1.03)
  Somnolence - Baseline | 1.0 (0.92)
  Somnolence - Week 12/EW | 0.5 (0.62)
  Somnolence - Change from Baseline | -0.5 (0.97)

7. Secondary Outcome: Change From Baseline at Week 12/Early Withdrawal (EW) in Johns Hopkins Restless Leg Syndrome Quality of Life Questionnaire (RLSQOL) on the Overall Life Impact Score
Description: The RLSQOL scale consists of 18 items, 13 of which are scored on a 5-point scale. Ten of the items can be summed to the overall life impact score, which can be transformed to a 0-100 score. Mild = 84.48, Moderate = 62.93, or Severe = 37.47
Time Frame: Baseline and Week 12/EW
Population: Full Analysis Set(FAS)
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 33
Points on a scale
  RLSQOL Overall Life Impact Score - Baseline | 65.29 (14.499)
  RLSQOL Overall Life Impact Score - Week 12 | 89.09 (13.431)
  Change from Baseline | 23.94 (16.759)

8. Primary Outcome: Haematology Clinical Lab Values Change From Baseline
Description: Standard units of measure vary. Therefore, Mean Change is represented in Standard Units: Hematocrit = SI unit of GSK; Hemoglobin = G/L; Platelet count, White Blood Cell count = GI/L; Red Blood Cell count = TI/L. n = number of subjects evaluated. EW = Early Withdrawal.
Time Frame: Baseline - Week 13 (Follow-up)
Population: Safety Population (Week 4 = 35 subjects, Week 8 = 32 subjects, Week 12 = 30 subjects, Week 12/EW = 33 subjects, Week 13 (Follow-up) = 35 subjects whose labs were evaluated).
Measure: Mean (Standard Deviation); unit: Varied Standard Units of Measure
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Varied Standard Units of Measure
  Hemoglobin (G/L) - week 4 | -1.2 (6.97)
  Hemoglobin (G/L) - week 8 | -2.7 (8.79)
  Hemoglobin (G/L) - week 12 | -1.0 (4.84)
  Hemoglobin (G/L) - week 12/EW | -0.8 (4.69)
  Hemoglobin (G/L)- week 13 | -2.2 (7.30)
  Hematocrit (SI) - week 4 | -0.0033 (0.01972)
  Hematocrit (SI) - week 8 | -0.0074 (0.02470)
  Hematocrit (SI) - week 12 | -0.0021 (0.01174)
  Hematocrit (SI) - week 12/EW | -0.0016 (0.01148)
  Hematocrit (SI) - week 13 | -0.0063 (0.01929)
  Platelet Count (GI/L) - week 4 | 14.5 (26.86)
  Platelet Count (GI/L) - week 8 | 11.7 (27.92)
  Platelet Count (GI/L) - week 12 | 8.5 (22.79)
  Platelet Count (GI/L) - week 12/EW | 8.8 (21.74)
  Platelet Count (GI/L) - week 13 | 10.7 (41.48)
  Red Blood Cell Count (TI/L) - week 4 | -0.043 (0.2139)
  Red Blood Cell Count (TI/L) - week 8 | -0.084 (0.2701)
  Red Blood Cell Count (TI/L) - week 12 | -0.015 (0.1469)
  Red Blood Cell Count (TI/L) - week 12/EW | -0.011 (0.1411)
  Red Blood Cell Count (TI/L) - week 13 | -0.050 (0.2140)
  White Blood Cell Count (GI/L) - week 4 | -0.191 (1.1655)
  White Blood Cell Count (GI/L) - week 8 | -0.268 (1.8694)
  White Blood Cell Count (GI/L) - week 12 | -0.577 (1.4972)
  White Blood Cell Count (GI/L) - week 12/EW | -0.516 (1.4407)
  White Blood Cell Count (GI/L) - week 13 | -0.624 (1.4914)

9. Primary Outcome: Blood Chemistry Clinical Lab Values Change From Baseline
Description: Mean Change in Standard Units of Measure: Albumin, Total Protein=G/L; Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Lactate Dehydrogenase, Creatine Phosphokinase, Gamma Glutamyl Transferase=IU/L; Total Bilirubin, Creatinine=UMOL/L; Blood Urea Nitrogen, Cholesterol, Chloride, Sodium, Potassium=MMOL/L; Prolactin=MCG/L
Time Frame: Baseline - Week 13 (Follow-up)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Varied Standard Units of Measure
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Varied Standard Units of Measure
  Albumin (G/L) - week 4 | -1.0 (2.35)
  Albumin (G/L) - week 8 | -1.4 (2.64)
  Albumin (G/L) - week 12 | -0.7 (2.34)
  Albumin (G/L) - week 12/EW | -0.6 (2.28)
  Albumin (G/L) - week 13 | -1.3 (2.33)
  Alkaline Phosphatase (IU/L) - week 4 | 5.2 (30.53)
  Alkaline Phosphatase (IU/L) - week 8 | 4.2 (26.94)
  Alkaline Phosphatase (IU/L) - week 12 | 13.2 (29.35)
  Alkaline Phosphatase (IU/L) - week 12/EW | 13.4 (28.52)
  Alkaline Phosphatase (IU/L) - week 13 | 16.0 (36.45)
  Alanine Amino Transferase (IU/L) - week 4 | -0.3 (3.80)
  Alanine Amino Transferase (IU/L) - week 8 | -0.7 (5.08)
  Alanine Amino Transferase (IU/L) - week 12 | 1.7 (4.66)
  Alanine Amino Transferase - week 12/EW | 1.8 (4.56)
  Alanine Amino Transferase - week 13 | 1.4 (6.36)
  Aspartate Amino Transferase(IU/L) - week 4 | 0.4 (4.55)
  Aspartate Amino Transferase (IU/L) - week 8 | -0.2 (4.07)
  Aspartate Amino Transferase (IU/L) - week 12 | 1.3 (4.57)
  Aspartate Amino Transferase (IU/L) - week 12/EW | 1.5 (4.51)
  Aspartate Amino Transferase (IU/L) - week 13 | 0.6 (4.35)
  Total Bilirubin (UMOL/L) - week 4 | 0.147 (3.1686)
  Total Bilirubin (UMOL/L) - week 8 | -0.588 (2.5180)
  Total Bilirubin (UMOL/L) - week 12 | 0.513 (3.4244)
  Total Bilirubin (UMOL/L) - week 12/EW | 0.311 (3.3513)
  Total Bilirubin (UMOL/L) - week 13 | -1.173 (3.7959)
  Blood Urea Nitrogen (MMOL/L) - week 4 | -0.14382 (1.079245)
  Blood Urea Nitrogen (MMOL/L) - week 8 | -0.06024 (0.862798)
  Blood Urea Nitrogen (MMOL/L) - week 12 | 0.25704 (1.076664)
  Blood Urea Nitrogen (MMOL/L) - week 12/EW | 0.30399 (1.043047)
  Blood Urea Nitrogen (MMOL/L) - week 13 | 0.32334 (0.974457)
  Cholesterol (MMOL/L) - week 4 | -0.093835 (0.5322345)
  Cholesterol (MMOL/L) - week 8 | -0.190717 (0.4337538)
  Cholesterol (MMOL/L) - week 12 | 0.151712 (0.5674075)
  Cholesterol (MMOL/L) - week 12/EW | 0.146540 (0.5494743)
  Cholesterol - week 13 | -0.107873 (0.5638668)
  Chloride(MMOL/L) - week 4 | 0.1 (1.78)
  Chloride (MMOL/L) - week 8 | 0.3 (2.07)
  Chloride (MMOL/L) - week 12 | -0.3 (1.81)
  Chloride (MMOL/L) - week 12/EW | -0.2 (1.92)
  Chloride (MMOL/L) - week 13 | -0.1 (2.30)
  Lactate Dehydrogenase (IU/L) - week 4 | 0.3 (22.02)
  Lactate Dehydrogenase (IU/L) - week 8 | -1.3 (16.74)
  Lactate Dehydrogenase (IU/L) - week 12 | 2.0 (25.96)
  Lactate Dehydrogenase (IU/L) - week 12/EW | 2.7 (25.06)
  Lactate Dehydrogenase (IU/L) - week 13 | -2.2 (18.78)
  Sodium (MMOL/L) - week 4 | -0.4 (1.37)
  Sodium (MMOL/L) - week 8 | -0.2 (1.36)
  Sodium (MMOL/L) - week 12 | 0.0 (1.11)
  Sodium (MMOL/L) - week 12/EW | -0.0 (1.07)
  Sodium (MMOL/L) - week 13 | -0.2 (1.29)
  Prolactin (MCG/L) - week 4 | 0.80 (7.003)
  Prolactin (MCG/L) - week 8 | 0.51 (7.229)
  Prolactin (MCG/L) - week 12 | 0.20 (6.770)
  Prolactin (MCG/L) - week 12/EW | 0.22 (6.466)
  Prolactin (MCG/L) - week 13 | 1.14 (7.144)
  Total Protein (G/L) - week 4 | -1.1 (3.73)
  Total Protein (G/L) - week 8 | -1.7 (4.03)
  Total Protein (G/L) - week 12 | -0.8 (3.32)
  Total Protein (G/L) - week 12/EW | -0.8 (3.20)
  Total Protein (G/L) - week 13 | -2.2 (3.45)
  Creatine Phosphokinase (IU/L) - week 4 | 72.3 (533.72)
  Creatine Phosphokinase (IU/L) - week 8 | -15.8 (100.86)
  Creatine Phosphokinase (IU/L) - week 12 | -0.6 (115.92)
  Creatine Phosphokinase (IU/L) - week 12/EW | -0.2 (110.40)
  Creatine Phosphokinase (IU/L) - week 13 | -1.9 (124.63)
  Creatinine (UMOL/L) - week 4 | 1.3134 (4.76710)
  Creatinine (UMOL/L) - week 8 | 0.5801 (7.23972)
  Creatinine (UMOL/L) - week 12 | 1.0019 (4.73343)
  Creatinine (UMOL/L) - week 12/EW | 1.0447 (4.60113)
  Creatinine (UMOL/L) - week 13 | 1.6417 (4.96904)
  Gamma Glutamyl Transferase (IU/L) - week 4 | 1.5 (17.56)
  Gamma Glutamyl Transferase (IU/L) - week 8 | -1.4 (11.68)
  Gamma Glutamyl Transferase (IU/L) - week 12 | 1.9 (14.56)
  Gamma Glutamyl Transferase (IU/L) - week 12/EW | 2.6 (14.26)
  Gamma Glutamyl Tranferase (IU/L) - week 13 | 0.1 (10.10)
  Potassium (MMOL/L) - week 4 | 0.07 (0.280)
  Potassium (MMOL/L) - week 8 | 0.05 (0.363)
  Potassium (MMOL/L) - week 12 | 0.09 (0.305)
  Potassium (MMOL/L) - week 12/EW | 0.10 (0.293)
  Potassium (MMOL/L) - week 13 | 0.06 (0.308)

10. Primary Outcome: Urinalysis Clinical Lab Values
Description: Dipstick test values: Neg Value, Trace, +1, +2, +3. No subjects tested higher than +3.
Time Frame: Baseline - Week 13 (Follow-up)
Population: Safety Population (Baseline, Week 4 = 35 subjects, Week 8 = 32 subjects, Week 12 = 30 subjects, Week 12/EW = 33 subjects, Week 13 [Follow-up] = 35 subjects evaluated).
Measure: Number; unit: Participants
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Participants
  Urine Urobilinogen - Baseline: Neg Value | 0
  Urine Urobilinogen - Baseline: Trace | 35
  Urine Urobilinogen - Baseline: +1 | 0
  Urine Urobilinogen - Baseline: +2 | 0
  Urine Urobilinogen - Baseline: +3 | 0
  Urine Urobilinogen - week 4: Neg Value | 0
  Urine Urobilinogen - week 4: Trace | 35
  Urine Urobilinogen - week 4: +1 | 0
  Urine Urobilinogen - week 4: +2 | 0
  Urine Urobilinogen - week 4: +3 | 0
  Urine Urobilinogen - week 8: Neg Value | 0
  Urine Urobilinogen - week 8: Trace | 32
  Urine Urobilinogen - week 8: +1 | 0
  Urine Urobilinogen - week 8: +2 | 0
  Urine Urobilinogen - week 8: +3 | 0
  Urine Urobilinogen - week 12: Neg Value | 0
  Urine Urobilinogen - week 12: Trace | 30
  Urine Urobilinogen - week 12: +1 | 0
  Urine Urobilinogen - week 12: +2 | 0
  Urine Urobilinogen - week 12: +3 | 0
  Urine Urobilinogen - week 12/EW: Neg Value | 0
  Urine Urobilinogen - week 12/EW: Trace | 33
  Urine Urobilinogen - week 12/EW: +1 | 0
  Urine Urobilinogen - week 12/EW: +2 | 0
  Urine Urobilinogen - week 12/EW: +3 | 0
  Urine Urobilinogen - week 13: Neg Value | 0
  Urine Urobilinogen - week 13: Trace | 35
  Urine Urobilinogen - week 13: +1 | 0
  Urine Urobilinogen - week 13: +2 | 0
  Urine Urobilinogen - week 13: +3 | 0
  Urine Protein - Baseline: Neg Value | 34
  Urine Protein - Baseline: Trace | 1
  Urine Protein - Baseline: +1 | 0
  Urine Protein - Baseline: +2 | 0
  Urine Protein - Baseline: +3 | 0
  Urine Protein - Week 4: Neg Value | 35
  Urine Protein - Week 4: Trace | 0
  Urine Protein - Week 4: +1 | 0
  Urine Protein - Week 4: +2 | 0
  Urine Protein - Week 4: +3 | 0
  Urine Protein - Week 8: Neg Value | 31
  Urine Protein - Week 8: Trace | 1
  Urine Protein - Week 8: +1 | 0
  Urine Protein - Week 8: +2 | 0
  Urine Protein - Week 8: +3 | 0
  Urine Protein - Week 12: Neg Value | 30
  Urine Protein - Week 12: Trace | 0
  Urine Protein - Week 12: +1 | 0
  Urine Protein - Week 12: +2 | 0
  Urine Protein - Week 12: +3 | 0
  Urine Protein - Week 12/EW: Neg Value | 33
  Urine Protein - Week 12/EW: Trace | 0
  Urine Protein - Week 12/EW: +1 | 0
  Urine Protein - Week 12/EW: +2 | 0
  Urine Protein - Week 12/EW: +3 | 0
  Urine Protein - Week 13: Neg Value | 35
  Urine Protein - Week 13: Trace | 0
  Urine Protein - Week 13: +1 | 0
  Urine Protein - Week 13: +2 | 0
  Urine Protein - Week 13: +3 | 0
  Urine Occult Blood - Baseline: Neg Value | 27
  Urine Occult Blood - Baseline: Trace | 5
  Urine Occult Blood - Baseline: +1 | 3
  Urine Occult Blood - Baseline: +2 | 0
  Urine Occult Blood - Baseline: +3 | 0
  Urine Occult Blood - Week 4: Neg Value | 20
  Urine Occult Blood - Week 4: Trace | 7
  Urine Occult Blood - Week 4: +1 | 6
  Urine Occult Blood - Week 4: +2 | 2
  Urine Occult Blood - Week 4: +3 | 0
  Urine Occult Blood - Week 8: Neg Value | 25
  Urine Occult Blood - Week 8: Trace | 3
  Urine Occult Blood - Week 8: +1 | 3
  Urine Occult Blood - Week 8: +2 | 0
  Urine Occult Blood - Week 8: +3 | 1
  Urine Occult Blood - Week 12: Neg Value | 23
  Urine Occult Blood - Week 12: Trace | 4
  Urine Occult Blood - Week 12: +1 | 2
  Urine Occult Blood - Week 12: +2 | 1
  Urine Occult Blood - Week 12: +3 | 0
  Urine Occult Blood - Week 12/EW: Neg Value | 25
  Urine Occult Blood - Week 12/EW: Trace | 5
  Urine Occult Blood - Week 12/EW: +1 | 2
  Urine Occult Blood - Week 12/EW: +2 | 1
  Urine Occult Blood - Week 12/EW: +3 | 0
  Urine Occult Blood - Week 13: Neg Value | 26
  Urine Occult Blood - Week 13: Trace | 3
  Urine Occult Blood - Week 13: +1 | 6
  Urine Occult Blood - Week 13: +2 | 0
  Urine Occult Blood - Week 13: +3 | 0
  Urine Glucose - Baseline: Neg Value | 35
  Urine Glucose - Baseline: Trace | 0
  Urine Glucose - Baseline: +1 | 0
  Urine Glucose - Baseline: +2 | 0
  Urine Glucose - Baseline: +3 | 0
  Urine Glucose - Week 4: Neg Value | 34
  Urine Glucose - Week 4: Trace | 0
  Urine Glucose - Week 4: +1 | 1
  Urine Glucose - Week 4: +2 | 0
  Urine Glucose - Week 4: +3 | 0
  Urine Glucose - Week 8: Neg Value | 31
  Urine Glucose - Week 8: Trace | 1
  Urine Glucose - Week 8: +1 | 0
  Urine Glucose - Week 8: +2 | 0
  Urine Glucose - Week 8: +3 | 0
  Urine Glucose - Week 12: Neg Value | 29
  Urine Glucose - Week 12: Trace | 1
  Urine Glucose - Week 12: +1 | 0
  Urine Glucose - Week 12: +2 | 0
  Urine Glucose - Week 12: +3 | 0
  Urine Glucose - Week 12/EW: Neg Value | 32
  Urine Glucose - Week 12/EW: Trace | 1
  Urine Glucose - Week 12/EW: +1 | 0
  Urine Glucose - Week 12/EW: +2 | 0
  Urine Glucose - Week 12/EW: +3 | 0
  Urine Glucose - Week 13: Neg Value | 35
  Urine Glucose - Week 13: Trace | 0
  Urine Glucose - Week 13: +1 | 0
  Urine Glucose - Week 13: +2 | 0
  Urine Glucose - Week 13: +3 | 0

11. Primary Outcome: 12-Lead Electrocardiogram (ECG) Findings Transitions From Baseline
Description: Baseline Finding/Time Period Finding. Abbreviations: N = normal; A = abnormal; CS = clinically significant; NCS = not clinically significant. Options include N/N, N/ANCS, N/ACS, ANCS/N, ANCS/ANCS, ANCS/ACS, ACS/N, ACS/ANCS, and ACS/ACS.
Time Frame: Baseline, Week 4, 8, 12, 13 (Follow-up)
Population: Safety Population - (Baseline = 35 subjects, Week 4 = 33 subjects, Week 8 = 31 subjects, Week 12/EW = 33 subjects and Week 13 [Follow-up] = 35 subjects evaluated).
Measure: Number; unit: Participants
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Participants
  Baseline: N; Baseline: N | 29
  Baseline: N; Baseline: ANCS | 0
  Baseline: N; Baseline: ACS | 0
  Baseline: ANCS; Baseline: N | 0
  Baseline: ANCS; Baseline: ANCS | 5
  Baseline: ANCS; Baseline: ACS | 0
  Baseline: ACS; Baseline: N | 0
  Baseline; ACS; Baseline: ANCS | 0
  Baseline: ACS ; Baseline: ACS | 1
  Baseline: N; Week 4: N | 27
  Baseline: N; Week 4: ANCS | 1
  Baseline: N; Week 4: ACS | 0
  Baseline: ANCS; Week 4: N | 2
  Baseline: ANCS; Week 4: ANCS | 1
  Baseline: ANCS; Week 4: ACS | 1
  Baseline: ACS; Week 4: N | 0
  Baseline: ACS; Week 4: ANCS | 0
  Baseline: ACS; Week 4: ACS | 1
  Baseline: N; Week 8: N | 24
  Baseline: N; Week 8: ANCS | 2
  Baseline: N; Week 8: ACS | 0
  Baseline: ANCS; Week 8: N | 2
  Baseline: ANCS; Week 8: ANCS | 1
  Baseline: ANCS; Week 8: ACS | 1
  Baseline: ACS; Week 8: N | 0
  Baseline: ACS; Week 8: ANCS | 1
  Baseline: ACS; Week 8: ACS | 0
  Baseline: N; Week 12/EW: N | 27
  Baseline: N; Week 12/EW: ANCS | 0
  Baseline: N; Week 12/EW: ACS | 0
  Baseline: ANCS; Week 12/EW: N | 4
  Baseline: ANCS; Week 12/EW: ANCS | 0
  Baseline: ANCS; Week 12/EW: ACS | 1
  Baseline: ACS; Week 12/EW: N | 0
  Baseline: ACS; Week 12/EW: ANCS | 0
  Baseline: ACS; Week 12/EW: ACS | 1
  Baseline: N; Week 13: N | 27
  Baseline: N; Week 13: ANCS | 2
  Baseline: N; Week 13: ACS | 0
  Baseline: ANCS; Week 13: N | 2
  Baseline: ANCS; Week 13: ANCS | 2
  Baseline: ANCS; Week 13: ACS | 1
  Baseline: ACS; Week 13: N | 0
  Baseline: ACS; Week 13: ANCS | 0
  Baseline: ACS; Week 13: ACS | 1

12. Primary Outcome: Vital Signs and Body Weight Change From Baseline
Description: Units of Measure Vary: Weight = kg; Semi-supine and Standing Systolic and Diastolic BP = mmHg; Semi-supine and Standing Pulse Rate = bpm; EW = early withdrawal; Semi-supine = lying down; Orthostatic = lying, sitting, and standing.
Time Frame: Baseline to Week 12/EW
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Varied Standard Units of Measure
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 33
Varied Standard Units of Measure
  Weight (Kg) | 0.5 (1.33)
  Semi-Supine Systolic BP (mmHg) | 2.7 (10.68)
  Semi-Supine Diastolic BP (mmHg) | 2.6 (7.25)
  Semi-Supine Pulse Rate (bpm) | 0.8 (9.11)
  Standing Systolic BP (mmHg) | -0.7 (10.86)
  Standing Diastolic BP (mmHg) | 0.8 (7.64)
  Standing Pulse Rate (bpm) | 1.1 (9.94)
  Orthostatic Systolic BP (mmHg) | -1.5 (8.50)
  Orthostatic Diastolic BP (mmHg) | 4.3 (5.58)
  Orthostatic Pulse Rate (bpm) | 9.2 (9.15)

13. Secondary Outcome: Change From Baseline at Week 12/Early Withdrawal (EW) in Profile of Mood Status (POMS)
Description: The POMS Standard form contains 65 items (0-232). The respondent rates each item on a 5-point scale, ranging from "Not at all (0)" to "Extremely (4)." The assessment measures six identified mood factors:
  * Tension-Anxiety
  * Depression-Dejection
  * Anger-Hostility
  * Vigor-Activity
  * Fatigue-Inertia
  * Confusion-Bewilderment
Time Frame: Baseline and Week 12/EW
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 33
Points on a scale
  POMS - Baseline | 59.2 (21.59)
  POMS - Week 12/EW | 48.0 (18.69)
  Change from Baseline | -10.4 (14.46)

14. Secondary Outcome: Change From Baseline at Week 12/Early Withdrawal (EW) in Hospital Anxiety and Depression Scale (HADS)
Description: Self screening questionnaire that requires the first response to questions. Questionnaire consists of 14 questions, seven for anxiety "0-21" and seven for depression "0-21". Questions are answered on a four point scale from 0-3; Items 1, 3, 5, 6, 8, 10, 11, and 13 are reversed for summation.
Time Frame: Baseline - Week 12/EW
Population: FAS: Subpopulation: HADS Anxiety population, N = 15; HADS Depression population, N = 31. Patients in the FAS population who also have a baseline anxiety domain score of 8 or greater and patients with a baseline depression domain score of 8 or greater will be included in the HADS Anxiety Population and the HADS Depression Population, respectively.
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
Points on a scale
  Anxiety-HADS Anxiety Population - Baseline | 9.3 (1.50)
  Anxiety-HADS Anxiety Population - Week 12/EW | 7.7 (2.39)
  Change from Baseline for Anxiety Population | -1.8 (2.58)
  Depression-HADS Depression Population -Baseline | 9.7 (1.42)
  Depression-HADS Depression Population-Week 12/EW | 9.5 (1.57)
  Change from Baseline for Depression Population | -0.1 (1.77)

15. Secondary Outcome: Pharmacokinetic Analysis: Plasma Concentrations of SK&F101468, an Unchanged Form of Ropinirole.
Description: Plasma samples taken at 24 hours after dosing had been administered for 3 days or longer. This was repeated if the dose was escalated. Lower Limits of Quantitation (LLQ) for SK&101468 = 20 pg/mL. The lowest concentration of analyte can be measured with established acceptable accuracy and precision.
Time Frame: Weeks 1-12
Population: Pharmacokinetic (PK) Population: subjects who underwent blood sampling for measuring the trough plasma drug concentrations, excluding those who did not fulfill inclusion criteria, those who were considered to affect the evaluation of the PK research due to drug incompliance or other protocol violation.
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
picograms/mL
  35 subjects who received 0.5 mg of Study drug | 310.01 (188.460)
  27subjects who received 1 mg of Study drug | 500.97 (293.344)
  11 subjects who received 2 mg of Study drug | 968.36 (696.327)
  2 subjects who received 3 mg of Study drug | 1294.55 (442.861)
  2 subjects who received 4 mg of Study drug | 1198.10 (362.463)

16. Secondary Outcome: Pharmacokinetic Analysis: Plasma Concentrations of SK&F104557, a Circulating Metabolite of Ropinirole.
Description: Plasma samples taken at 24 hours after dosing had been administered for 3 days or longer. This was repeated if the dose was escalated. Lower Limits of Quantitation (LLQ) for SK&104557 = 20 pg/mL. The lowest concentration of analyte can be measured with established acceptable accuracy and precision.
Time Frame: Weeks 1 -12
Population: PK Population
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
picograms/mL
  35 subjects who received 0.5 mg of Study drug | 324.65 (134.576)
  27 subjects who received 1 mg of Study drug | 615.91 (259.145)
  11 subjects who received 2 mg of Study drug | 1320.31 (523.622)
  2 subjects who received 3 mg of Study drug | 1666.65 (325.764)
  2 subjects who received 4 mg of Study drug | 2541.95 (198.202)

17. Secondary Outcome: Pharmacokinetic Analysis: Plasma Concentrations of SK&F89124, a Circulating Metabolite of Ropinirole.
Description: Plasma samples taken at 24 hours after dosing had been administered for 3 days or longer. This was repeated if the dose was escalated. Lower Limits of Quantitation (LLQ) for SK&89124 = 20 pg/mL. The lowest concentration of analyte can be measured with established acceptable accuracy and precision.
Time Frame: Weeks 1-12
Population: PK Population
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Ropinirole CR-RLS
Number analyzed (Participants) | 35
picograms/mL
  2 subjects who received 0.5 mg of Study drug | 22.45 (3.465)
  11 subjects who received 1 mg of Study drug | 30.37 (10.227)
  11 subjects who received 2 mg of Study drug | 42.75 (17.286)
  2 subjects who received 3 mg of Study drug | 46.80 (8.202)
  2 subjects who received 4 mg of Study drug | 72.05 (2.051)

ADVERSE EVENTS:
Arm/Group | Ropinirole CR-RLS
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 33/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole CR-RLS (N=35)
Nausea (Gastrointestinal disorders) | 15
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 12
Somnolence (Psychiatric disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Dizziness (General disorders) | 3
Hypersomnia (Psychiatric disorders) | 3
Anemia (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Gingivitis (Infections and infestations) | 2
Stomach Discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal Pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood urine present (Investigations) | 1
Chillblains (Injury, poisoning and procedural complications) | 1
Cold Sweat (Skin and subcutaneous tissue disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Irritability (General disorders) | 1
Local Swelling (General disorders) | 1
Malaise (General disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Motion sickness (Ear and labyrinth disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Palpitations (Cardiac disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pyrexia (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 1
Tenosynovitis (Skin and subcutaneous tissue disorders) | 1
Tension headache (Nervous system disorders) | 1
Thirst (General disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Upper Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Vertebral injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of the multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.